CLINICAL TRIAL: NCT02234180
Title: Randomized Phase II Double Blind Study of Adjuvant Regorafenib vs Placebo in Patients With Node Positive Esophageal Cancer That Completed Pre-operative Therapy
Brief Title: Regorafenib in Treating Patients With Locally Advanced Cancer of the Esophagus or Gastroesophageal Junction Who Have Completed Chemoradiation Therapy and Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RU021212I; NCI-2015-01699 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2014-01962; RU021212I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Stage IIB Esophageal Adenocarcinoma; Stage IIIA Esophageal Adenocarcinoma; Stage IIIB Esophageal Adenocarcinoma; Stage IIIC Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (regorafenib) (Experimental): Within 6-12 weeks after surgery, patients receive regorafenib PO QD on days 1-21. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Regorafenib
- Arm II (placebo) (Placebo Comparator): Within 6-12 weeks after surgery, patients receive placebo PO QD on days 1-21. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; Stivarga
  Arms: Arm I (regorafenib)

SUMMARY:
This randomized phase II trial studies how well regorafenib works in treating patients with cancer of the esophagus or gastroesophageal junction that has spread from where it started to nearby tissue or lymph nodes and have completed chemoradiation therapy and surgery. Regorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the disease-free survival (DFS) for patients with resected esophageal and gastroesophageal (GE) junction adenocarcinoma treated with regorafenib vs. placebo in the adjuvant setting.

SECONDARY OBJECTIVES:

I. To compare the safety profile of adjuvant regorafenib vs. placebo in patients with locally advanced resectable esophageal and GE junction adenocarcinoma.

II. To compare the overall survival (OS) for patients with resected esophageal and GE junction adenocarcinoma treated with regorafenib vs. placebo in the adjuvant setting.

III. To compare the DFS in those patients that receive at least 1 cycle of therapy.

IV. To collect tumor samples for future genomic analysis to explore the biology of locally advanced esophageal and GE junction adenocarcinoma.

V. DFS will be compared between the arms from the time of surgery as well.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Within 6-12 weeks after surgery, patients receive regorafenib orally (PO) once daily (QD) on days 1-21.

ARM II: Within 6-12 weeks after surgery, patients receive placebo PO QD on days 1-21.

In both arms, courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years, and every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of node positive (any T stage N1-3) proximal esophageal, distal esophagus or gastroesophageal (GE) junction adenocarcinoma (Siewert I, II, or III) after completing preoperative chemoradiation and surgery; supporting pathology report sufficient for registration; available tumor tissue from endoscopic biopsies prior to preoperative chemotherapy (chemo)/radiation therapy (RT), and tumor from surgical specimens will be submitted to Academic and Community Cancer Research United (ACCRU), but not be required prior registration; Note: if tissue is depleted, patient will still be eligible after discussion with the physician
* Imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) =< 28 days of study registration negative for disease recurrence
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Lipase =< 1.5 x the ULN
* Serum creatinine =< 1.5 x the ULN
* International normalized ratio (INR)/partial thromboplastin time (PTT) =< 1.5 x ULN; Note-subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that their medication dose and INR/PTT are stable; close monitoring (day 1 of each cycle) is mandatory; if either of these values is above the therapeutic range, the doses should be modified and the assessments should be repeated weekly until they are stable
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Able to swallow and retain oral medications and begin therapy within 6 to 12 weeks post-surgery
* Provide blood samples for the mandatory correlative research purposes

Exclusion Criteria:

* Presence of metastatic or recurrent disease
* R1 or R2 resection
* Patients who have not recovered from serious adverse events (as determined by treating doctor of medicine [MD]) related to surgery
* Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg on repeated measurement) despite optimal medical management per physician discretion
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > class II
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Unstable angina (anginal symptoms at rest), new-onset angina < 3 months before randomization, or myocardial infarction within 6 months before randomization
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event >= National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4 grade 3 =< 4 weeks prior to registration
* Prior cancers < 3 years, with the exception of in-situ cervical cancer, low grade prostate cancer and basal or squamous cell skin cancers
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism =< 6 months prior to registration
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); use of strong or moderate inhibitors are prohibited =< 7 days to registration
* Receiving any medications or substances that are inducers of CYP3A4; use of inducers are prohibited =< 7 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Janjigian, Principal Investigator — Academic and Community Cancer Research United
Locations (10):
- United States (10):
  - Carle Cancer Center, Urbana, Illinois
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Regorafenib): Within 6-12 weeks after surgery, patients will receive regorafenib PO QD on days 1-21. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
- Arm II (Placebo): Within 6-12 weeks after surgery, patients will receive placebo PO QD on days 1-21. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Regorafenib) | Arm II (Placebo)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 1 patient was registered to the placebo arm. Due to protected health information, listing only 1 patient's results is contraindicated.
Groups:
- Arm I/II (Regorafenib/Placebo): Within 6-12 weeks after surgery, patients receive regorafenib OR placebo PO QD on days 1-21. Courses repeat every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I/II (Regorafenib/Placebo)
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 54.0 [53.0 to 58.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: Disease free survival (DFS) is defined as the time from randomization to the first of either disease recurrence or death from any cause. The distribution of DFS will be estimated using the Kaplan Meier method.
Time Frame: Time from randomization to the first of either disease recurrence or death from any cause, assessed up to 1 year and 10 months
Population: Only 1 patient was registered to the placebo arm. Due to protected health information, listing only 1 patient's results is contraindicated. The data below is descriptive and shouldn't be trusted because of the small sample size.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I/II (Regorafenib/Placebo)
Number analyzed (Participants) | 3
months | 4.83 [2.27 to 9.89]

2. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 1 year and 10 months
Population: as for outcome 1
Measure: Number; unit: percentage of grade 3+ AEs
Arm/Group | Arm I/II (Regorafenib/Placebo)
Number analyzed (Participants) | 3
percentage of grade 3+ AEs | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from randomization to death due to any cause.
Time Frame: Time from randomization to death due to any cause, assessed up to 1 year and 10 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I/II (Regorafenib/Placebo)
Number analyzed (Participants) | 3
months | NA [NA to NA] — No OS events observed among the patients, thus no OS median and 95% confidence interval is available.

ADVERSE EVENTS:
Time Frame: Up to 1 year and 10 months
Description: The descriptions & grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation & scientific analysis & is a single MedDRA Lowest Level Term (LLT). Only 1 patient was registered to the placebo arm. Due to protected health information, listing only 1 patient's results is contraindicated.
Arm/Group | Arm I/II (Regorafenib/Placebo)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I/II (Regorafenib/Placebo) (N=3)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I/II (Regorafenib/Placebo) (N=3)
Diarrhea (Gastrointestinal disorders) | 2 (6)
Vomiting (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (7)
Hypertension (Vascular disorders) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No